CLINICAL TRIAL: NCT07164040
Title: Fluorescence Visualization and Image Quality Evaluation of Digital Visualization During Standard of Care Procedure in the Cerebral Vascular Area as Well as Blood Flow During Plastic and Reconstructive Surgery (PRS) (Leica GLOW800)
Brief Title: Leica Microsystems Sponsored Study to Collect and Confirm Clinical Data on the Performance of the GLOW800 Device When Used in Accordance With Its Intended Use.
Acronym: IMED-GLOW800
Status: Recruiting | Type: Observational
Sponsor: Leica Microsystems (Schweiz) AG (Industry)
Responsible Party: Sponsor
Other Study IDs: GLOW800-PMCFSTUDYPLAN-202501
Record Dates: First submitted 2025-08-15; First posted 2025-09-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Reconstructive Surgical Procedures; Plastic Surgery; Vascular Surgical Procedure; Cerebrovascular Disorder
Keywords: GLOW800; Indocyanine-green (ICG); Near Infrared; plastic and reconstructive surgery; ARveo8X; Surgical Microscope; Fluorescence imaging; Cerebrovascular surgery; Intraoperative visualization; Post-market clinical follow-up (PMCF); Image quality assessment; 3D visualization; Heads-up surgery; Vascular imaging; Digital surgical workflow
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GLOW800
  Interventions: Device: The GLOW800, a non-contact, non-invasive device, allows the surgical microscope ARveo 8 and ARveo 8X to produce excitation light and resolve fluorescence emission from the fluorescent agent ICG

INTERVENTIONS:
Device: The GLOW800, a non-contact, non-invasive device, allows the surgical microscope ARveo 8 and ARveo 8X to produce excitation light and resolve fluorescence emission from the fluorescent agent ICG — When activating the GLOW800 mode, the white light illumination of the Leica microscope stand is extended to InfraRed (IR), to excite the fluorophore (ICG). The technology provides ergonomic advantages as the user can maintain an upright posture while observing the surgical field. To excite the fluorophore, ICG dye is illuminated with light at its excitation wavelength band around 750 - 800nm. GLOW800 utilizes a 400w xenon illumination light source integrated as a standard component within the compatible Surgical Operating Microscope (SOM) stand. Activation of the GLOW800 mode extends the white light illumination of the SOM to the infrared (IR) spectral range using a suitable filter placed in the compatible SOM's standard filter wheel for the excitation of the ICG. Each patient enrolled in this study will undergo standard of care for the surgical procedure. No deviations to the standard of care will occur in the execution of this study.

SUMMARY:
This post-market clinical follow-up (PMCF) study aims to confirm the safety and performance of the GLOW800 surgical microscope accessory when used in conjunction with the ARveo8x surgical microscope. The study evaluates fluorescence visualization and image quality during standard surgical procedures in the cerebral vascular area and plastic and reconstructive surgery. It is a non-interventional, observational study conducted in routine care settings across multiple European sites.

DETAILED DESCRIPTION:
The IMED-GLOW800 study is designed to collect clinical data on the GLOW800 device, a CE-marked surgical microscope accessory developed by Leica Microsystems. The device enables enhanced intraoperative visualization of blood flow using Indocyanine Green (ICG) fluorescence, integrated into the surgical field in real-time with stereoscopic depth perception.

Traditional ICG-guided surgery often requires switching between anatomical and fluorescence views, which can interrupt surgical workflow. GLOW800 overcomes this limitation by digitally overlaying fluorescence signals onto the anatomical view, improving surgical decision-making and workflow efficiency.

The study will enroll 31 patients across at least two sites in the European Economic Area (EEA) and Switzerland. Eligible patients will undergo standard surgical procedures in the cerebral vascular area or plastic and reconstructive surgery. The study does not involve additional invasive procedures and is conducted entirely within the scope of routine care.

The primary objective is to assess the performance of GLOW800 in terms of fluorescence visibility and image quality. Secondary objectives include evaluating the continued safety of the device. Data will be collected using structured questionnaires completed by surgeons during and after surgery, along with video recordings captured by the microscope.

Endpoints include:

Primary: Fluorescence visibility (monochrome and pseudo-color), anatomical and fluorescence observations, vessel architecture, blood flow, capillary transition, drainage, stereoscopic perception, resolution, latency, and real-time blood flow visibility.

Secondary: Safety indicators such as dizziness, surgical interruptions, injuries, sterility breaches, and tissue burns.

The study duration is estimated at 5-6 months from first patient enrollment to completion. Each patient will participate in a single surgical procedure with no follow-up required.

Data will be pseudonymized and managed in compliance with GDPR and ISO 14155:2020. The study is sponsored by Leica Microsystems (Schweiz) AG and will be monitored according to standard clinical research practices.

The results will contribute to ongoing post-market surveillance and may support regulatory submissions, scientific publications, and future product development.

ELIGIBILITY:
Inclusion Criteria:

Candidates for the study must be appropriate patients for surgical interventions in the cerebral vascular area or for plastic and reconstructive surgery and have to fulfil all of the following inclusion criteria to be eligible for the recruitment of the study.

1. Participants must be 18 years of age or older at the time of signing the informed consent.
2. Participants must have a condition requiring surgical intervention in the cerebral vascular area as well as during plastic and reconstructive surgery.
3. The Indocyanine Green (ICG) cyanine dye is administered as a contrast agent per instructions for use.
4. The participant or their legal representative must understand the study and have voluntarily signed and dated the Informed Consent Form, which has been approved by the Sponsor and the Ethics Committee for this study

Exclusion Criteria:

Candidates who meet any of the following exclusion criteria will not be eligible for recruitment in the study.

1. Known allergy to Indocyanine Green (ICG) cyanine dye.
2. Any uncontrolled systemic condition that may adversely affect the surgical outcome.
3. Patients holding United States citizenship.
4. Severe iodine-induced reactions to macromolecular iodine-containing compounds (e.g., iodinated contrast media, iodine-based antiseptics, or drugs like amiodarone), especially if the reaction involved anaphylaxis or respiratory compromise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population will include patients diagnosed with condition requiring surgical interventions in the cerebral vascular region as well as during plastic and reconstructive surgery and the patient needs to meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Fluorescence visibility. | Periprocedural
  Performance will be evaluated using Questionnaire, a structured Likert-scale survey completed by the operating surgeon during and after surgery.
  The questionnaire assesses:
  1. Perceived fluorescence visibility in monochrome view
  2. Perceived fluorescence visibility in pseudo color view
  3. Anatomical and fluorescence observation
  4. Fluorescence information given by Indocyanine Green (ICG)
  5. Fluorescence information about vessel architecture
  6. Fluorescence information about blood flow
  7. Fluorescence information about capillary transition
  8. Fluorescence information about drainage over venous blood vessels
  Each item is rated on a 5-point Likert scale:
  1. = Not available
  2. = Insufficient
  3. = Sufficient
  4. = Very good
  5. = Excellent Higher scores indicate better performance. The outcome is considered acceptable if all ratings are ≥3 (Sufficient or better).
Image quality | Periprocedural
  Performance will be evaluated using Questionnaire, a structured Likert-scale survey completed by the operating surgeon during and after surgery. The questionnaire assesses:
  1. Stereoscopic Perception (3D Depth perception)
  2. Resolution
  3. Latency
  Each item is rated on a 5-point Likert scale:
  1. = Not available
  2. = Insufficient
  3. = Sufficient
  4. = Very good
  5. = Excellent Higher scores indicate better performance. The outcome is considered acceptable if all ratings are ≥3 (Sufficient or better).
Anatomical background | Periprocedural
  Performance will be evaluated using Questionnaire A, a structured Likert-scale survey completed by the operating surgeon during and after surgery. The questionnaire assesses: The visibility of anatomical structures are rated.
  Each item is rated on a 5-point Likert scale:
  1. = Not available
  2. = Insufficient
  3. = Sufficient
  4. = Very good
  5. = Excellent Higher scores indicate better performance. The outcome is considered acceptable if all ratings are ≥3 (Sufficient or better.)
Visibility of real time vascular blood flow | Periprocedural
  Performance will be evaluated using Questionnaire A, a structured Likert-scale survey completed by the operating surgeon during and after surgery. The questionnaire assesses: Visibility of real-time vascular blood flow
  Each item is rated on a 5-point Likert scale:
  1. = Not available
  2. = Insufficient
  3. = Sufficient
  4. = Very good
  5. = Excellent Higher scores indicate better performance. The outcome is considered acceptable if all ratings are ≥3 (Sufficient or better).

SECONDARY OUTCOMES:
The secondary objectives of this Post-Market Clinical Follow-up (PMCF) study are to assess the continued safety of the device. | Postoperatively
  Safety will be evaluated using Questionnaire B, completed postoperatively by the surgical team. It captures:
  1. Dizziness through using digital 3D visualization
  2. Delayed, interrupted or hindered surgery due to different causes
  3. Occurred injuries to the patient
  4. Breach of sterility
  5. Any patient or user tissue burn event reported.
  Responses are binary:
  1. = Yes (event occurred)
  2. = No (event did not occur) Lower scores (2 = No) indicate better safety outcomes. The outcome is acceptable if no safety events are reported.

CONTACTS AND LOCATIONS:
Locations (3):
- Unidade Local de Saúde de São João, Porto, Portugal
- Hospital Germans Trias I Pujol, Barcelona, Spain
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication.
Supporting Information: Study Protocol, CSR